CLINICAL TRIAL: NCT06840808
Title: Using High Definition Transcranial Direct Current Stimulation to Treat Verbal Retrieval Deficits Secondary to Chronic Traumatic Brain Injury (HDtDCS-CTBI)
Brief Title: Treating Word Finding Difficulties in Traumatic Brain Injury With HD-tDCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU2022-0999/23-231; 23-231 (Other: The UNIVERSITY OF TEXAS AT DALLAS); STU2022-0999 (Other: UNIVERSITY OF TEXAS SOUTHWESTERN MEDICAL CENTER)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Cognitive Change; Word Finding Difficulty; Acquired Brain Injury
Keywords: electroencephalography; transcranial direct current stimulation; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic; Anomia; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 treatment arms: (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule.
  Additionally, after completing the initial active or sham treatment and 2-month follow-up testing sessions, all participants will be invited back for newly assigned treatment conditions, 20 minutes over 10 sessions and will be and re-evaluated at 2-months follow-up testing sessions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, assessors, and technicians interacting with participants will be blind to assigned conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active to Sham Transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive active stimulation. After completion of active stimulation, subjects will be assigned to sham stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation
- Sham to Active transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive sham stimulation. After completion of sham stimulation, subjects will be assigned to active stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Active Transcranial direct current stimulation — Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
Device: Sham Transcranial direct current stimulation — Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.

SUMMARY:
The purpose of the study is to test whether low level electric stimulation, called transcranial Direct Current Stimulation (tDCS), on the part of the brain (i.e., pre-supplementary motor area) thought to aid in memory will improve verbal retrieval in civilian (non-military, non-veteran) participants with histories of traumatic brain injuries. The primary outcome measures are neuropsychological assessments of verbal retrieval, and the secondary measures are neuropsychological assessments of other cognitive abilities and electroencephalography (EEG) measures. Additionally, the study will examine the degree to which baseline assessments of cognition, concussion history, structural brain imaging, and EEG predict responses to treatment over time, both on assessments administered within the intervention period and at follow-up.

DETAILED DESCRIPTION:
Using two treatment arms, the study will examine improvement of verbal retrieval and other cognitive deficits associated with remote traumatic brain injury by comparing (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule. Additionally, after completing the initial active or sham treatment and 2-month follow-up testing sessions, participants will be invited back for newly assigned treatment conditions, 20 minutes over 10 sessions and will be re-evaluated at 2-months follow-up testing sessions.

Civilians with histories of traumatic brain injuries and observed cognitive deficits will be randomly assigned to one of the two treatment arms (and re-assigned for the second round of intervention, as described above). Primary outcome verbal retrieval measures, secondary neuropsychological and electroencephalography (EEG) measures, and prescreening assessments for study concussion history and contraindications for treatment will be collected prior to being assigned to a treatment arm (i.e., baseline).

Primary outcome verbal retrieval measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected after treatment session 10 and one time following treatment competition (i.e., 2-months). For participants who complete the second round of intervention, primary outcome verbal memory measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected again after treatment session 10 and one time following competition of the second treatment (i.e., 2-months).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-85
* Traumatic brain injury more than a year prior to study participation
* Word finding difficulty since the brain injury
* Fluent in speaking and reading English.

Exclusion Criteria:

* Implanted/electronic device, such as a pacemaker, metallic cranial or intracranial implant (e.g., ventriculoperitoneal shunt), or a neurostimulator (e.g., vagus nerve stimulator, spinal stimulator, deep brain stimulator, etc.).
* Skull defects
* History of a psychological or neurological disorder, including, dementia of any type, epilepsy or other seizure disorders, post-traumatic stress disorder, brain tumor, present drug abuse, stroke, blood vessel abnormalities in the brain, Parkinson's disease, Huntington's disease, or multiple sclerosis.
* Inability to give informed consent
* Military personnel or Veteran
* Currently pregnant
* Not fluent English speaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Controlled Oral Word Association Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Control Word Association Test, including both letter and category fluency. Metric: Number of Correct Items Generated
The Boston Naming Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on The Boston Naming Test. Metric: Number of Correct Items Generated.
Rey Auditory Verbal Learning Test and alternative lists | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Rey Auditory Verbal Learning Test. Metric: Number of Total learning items and Correct Recalls.
The Delis Kaplan Color Word Interference Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Delis Kaplan Color Word Interference Test. Metric: Time to Name Items

SECONDARY OUTCOMES:
The Trail Making Test (Parts A & B) | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Trail Making Test (Parts A&B). Metric: Time to Solution
Digit Span Forward & Backward | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Digit Span Forward & Backward. Metric: Memory Span
Rey-Osterrieth Complex Figure Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Rey-Osterrieth Complex Figure Test scores. Metric: Score 0 to 36, the higher the better
The Digit Symbol Substitution Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Digit Symbol Substitution Test. Metric: Number of Items
Task-based electroencephalography (EEG) markers during a Go-NoGo task | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in EEG change on a Go-NoGo task with different levels of perceptual/semantic complexity. Metric: event-related potentials and time frequency changes.
Task-based electroencephalography (EEG) markers during a Semantic Object Memory Retrieval task | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in EEG change on a Semantic Object Retrieval task. Metric: event-related potentials and time frequency changes.

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, MD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will share data upon request.

REFERENCES:
- [Background] Motes MA, Spence JS, Yeatman K, Jones PM, Lutrell M, O'Hair R, Shakal S, DeLaRosa BL, To W, Vanneste S, Kraut MA, Hart J , Jr. High-Definition Transcranial Direct Current Stimulation to Improve Verbal Retrieval Deficits in Chronic Traumatic Brain Injury. J Neurotrauma. 2020 Jan 1;37(1):170-177. doi: 10.1089/neu.2018.6331. Epub 2019 Sep 3. PMID 31354040
- [Background] Chiang HS, Motes M, O'Hair R, Vanneste S, Kraut M, Hart J Jr. Baseline delayed verbal recall predicts response to high definition transcranial direct current stimulation targeting the superior medial frontal cortex. Neurosci Lett. 2021 Nov 1;764:136204. doi: 10.1016/j.neulet.2021.136204. Epub 2021 Sep 1. PMID 34478816
- [Background] Chiang HS, Motes M, Kraut M, Vanneste S, Hart J. High-definition transcranial direct current stimulation modulates theta response during a Go-NoGo task in traumatic brain injury. Clin Neurophysiol. 2022 Nov;143:36-47. doi: 10.1016/j.clinph.2022.08.015. Epub 2022 Aug 30. PMID 36108520